CLINICAL TRIAL: NCT03588949
Title: Role of Nutritional Support in Idiopathic Male Infertility: a Randomized Dietary Study
Brief Title: Role of Nutritional Support in Idiopathic Male Infertility
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: NATURAmedicatrix Sàrl (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: NATURAmedicatrix-FE-0001-M
Record Dates: First submitted 2018-06-26; First posted 2018-07-17 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2019-08

CONDITIONS: Infertility, Male
MeSH Terms: conditions — Infertility, Male | interventions — Dietary Supplements; Carnitine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Dietary Supplement (Experimental): Dietary Supplement with L-carnitine (FertilHom)
  Interventions: Dietary Supplement: Dietary Supplement with L-carnitine (FertilHom)
- Control Dietary Supplement (Placebo Comparator): Dietary Supplement with 50% RDA of beta-carotene
  Interventions: Dietary Supplement: Control Dietary Supplement

INTERVENTIONS:
Dietary Supplement: Dietary Supplement with L-carnitine (FertilHom) — 1 stick of the TDS (vitamins, trace elements with carnitine) will be given 1 time daily in the evening before meals for 6 months or until pregnancy, depending whatever comes first
  Arms: Active Dietary Supplement
Dietary Supplement: Control Dietary Supplement — 1 stick of the TDSwill be given 1 time daily in the evening before meals for 6 months or until pregnancy, depending whatever comes first
  Arms: Control Dietary Supplement

SUMMARY:
Approximately 100 males with idiopathic infertility and oligo- and/or astheno- and/or and/or teratozoospermia and fertile woman will take a Test dietary supplement (TDS), containing carnitine, vitamins and trace elements (active group) or carotene (control group) for 6 months (50 subjects in active and control groups). Before intake, and 2 and 4 months after the commencement of TDS, all males will have spermogram. After 6-month use of the TDS and during the 12th month of the study, couples will be screened for conception, pregnancy, and a newborn

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent form signed;
2. Age: 21-50;
3. Idiopathic male infertility;
4. Idiopathic oligo- and/or astheno- and/or teratozoospermia;
5. Stated availability throughout the study period and a mobile phone

Exclusion Criteria:

1. Allergy to any component of the dietary supplement;
2. Known genetic, anatomical, endocrine, inflammatory or traumatic testicular cause of male infertility;
3. Known genetic, anatomical, endocrine, inflammatory or traumatic testicular cause of female infertility;
4. Inflammatory bowel disease;
5. Known moderate to severe disease of any systems;
6. Known or suspected sexually transmitted diseases;
7. Alcohol or drug addiction of any couple counterpart as suspected by investigator;
8. Difficulty to comprehend study requirements as judged by investigator;
9. Use of any investigational product within the previous 3 months before entering the study;
10. Use of any drugs that stimulate or suppress spermatogenesis within previous 3 months

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-04-30 (Estimated)

PRIMARY OUTCOMES:
Rate of normalization of spermogram | 4 months
  None deviation found in spermogram

CONTACTS AND LOCATIONS:
Overall Officials: Marco Pietteur, Study Director — NATURAmedicatrix Sarl
Locations (1):
- MedianaStatistics, Lviv, Ukraine